CLINICAL TRIAL: NCT05077670
Title: Hybrid Characterization of Driver Sites During Atrial Fibrillation and Sinus Rhythm With CARTOFINDER and COHERENT Mapping
Brief Title: Hybrid Characterization of Driver Sites During Atrial Fibrillation and Sinus Rhythm
Acronym: Hybrid-AFMAP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundacion para la Innovacion en Biomedicina (FIBMED) (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Hybrid-AFMAP
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Catheter ablation; Rotors
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Study group: * LAA + LA Map in AF
  * Identify LAA connections and detect rotors with CartoFinder
  * Electrical cardioversion. Sinus rhythm restoration
  * Pacing from the coronary sinus at 300 and 600ms periods
  * Analyze COHERENT activation maps in sinus rhythm
  * Ablation as suggested by current clinical guidelines and the characteristics of the patient
  Interventions: Procedure: Pulmonary vein electrical isolation; Device: Atrial substrate mapping

INTERVENTIONS:
Procedure: Pulmonary vein electrical isolation — Electrical isolation of the pulmonary veins from the left atrium with cryoablation therapy.
  Other Names: Pulmonary veins ablation
Device: Atrial substrate mapping — Electro-anatomical maps will be performed with CARTO navigation system with multi-electrode catheters.
  Other Names: Electro-anatomical mapping

SUMMARY:
The primary objective of this study is twofold, first we aim to identify rotors in atrial fibrillation (AF) and analyze their relationship with the left atrium-left atrial appendage (LA-LAA) connections. Secondly, we will analyze the areas harboring rotors in SR to define the characteristics that describe the presence of rotors.

DETAILED DESCRIPTION:
The primary objective of this study is the identification of LA and LAA areas driving atrial fibrillation to study their relationship with LAA-LA connections and sinus rhythm (SR) analysis using the CartoFinder and COHERENT algorithms that CARTO V7 offers.

The CartoFinder tool will be able to determine the activation patterns of reentrant drivers (rotors) in the LA and LAA in AF. The characterization of areas harboring rotors could be performed with the COHERENT tool provided by CARTO V7 to determine the activation patterns during reentrant rhythms, and after sinus rhythm restoration it could be used to assess the conduction patterns at LA-LAA connections and driver sites identified with CartoFinder.

ELIGIBILITY:
Inclusion Criteria:

* Persistent atrial fibrillation
* The patient has signed the informed consent form
* No LAA previous ablation procedure
* No valvular disease
* LVEF ≥ 35% prior to recruitment
* Age ≥ 18 years

Exclusion Criteria:

* LVEF < 35 %
* Hyperthyroidism or hypothyroidism
* Mental or physical illness incapacitation
* Planned cardiac procedure
* Non-controlled hypertension
* Terminal renal failure or dialysis
* Class IV of the NYHA
* Age ≥ 75 years
* Life expectancy < 2 years
* Atrioventricular block
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include 50 patients. No statistical considerations were made to determine the sample size of this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
CartoFinder and COHERENT tools utility assessment | 2 years
  To evaluate the utility of CartoFinder and COHERENT tools in the identification of the mechanisms that maintain atrial fibrillation.

SECONDARY OUTCOMES:
Atrial fibrillation driver location analysis | 2 years
  Reentrant driver location relationship with lines of block, wavefront curvature, and slow conduction areas during SR pacing with success AF termination.

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Arenal, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón; Gonzalo R Ríos-Muñoz, MSc, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No